CLINICAL TRIAL: NCT04407416
Title: The Effectiveness of Breath Analysis Versus FIT for Colorectal Cancer Screening
Brief Title: VOCs vs FIT for Colorectal Cancer Screening
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Societa Italiana di Chirurgia ColoRettale (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 27/2020
Record Dates: First submitted 2020-05-22; First posted 2020-05-29 (Actual); Last update posted 2020-05-29 (Actual); Status verified 2020-05

CONDITIONS: Colorectal Cancer; Colorectal Polyp
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Healthy subjects (Active Comparator): The breath of all patients with positive FIT (fecal immunochemical test) but negative colonoscopy will be sampled using a breath sampler
  Interventions: Procedure: Breath sampling
- Colorectal Cancer patients (Active Comparator): The breath of all patients with positive FIT (fecal immunochemical test) and a colorectal cancer detected by colonoscopy will be sampled using a breath sampler
  Interventions: Procedure: Breath sampling
- Colonic Polyps patients (Active Comparator): The breath of all patients with positive FIT (fecal immunochemical test) and a colonic polyp detected by colonoscopy will be sampled using a breath sampler
  Interventions: Procedure: Breath sampling

INTERVENTIONS:
Procedure: Breath sampling — The breath of all subjects included will be sampled using a device able to capture the alveolar air and to fix it on carbon tubes, Then the tubes will be desorbed and analysed using gas chromatography

SUMMARY:
Endogenous breath VOCs (Volatile Organic Compounds) are present in various excreted biological materials (urine, blood, faeces an breath) and their analysis offers a possibility for cancer screening. Some of these VOCs are reversed in the venous blood stream and reach the lung alveoli where some of them are exhaled.

Colorectal cancer (CRC) is one of the commonest tumours and is an important cause of cancer-related mortality. Colonoscopy is the gold standard for the diagnosis of CRC.

Screening with fecal immunochemical test (FIT) is associated with a 13-18% CRC-mortality reduction.

Aim of the study To compare the reliability of this breath analysis with Immunochemically-based Fecal Occult Blood Test.

DETAILED DESCRIPTION:
Volatile organic compounds (VOCs) are low molecular weight (<1 kDa) compounds which represent the final products of cell metabolism. Their composition can be affected by several factors including diet, hormones, environment and the presence of diseases, in particular, cancer.

Endogenous breath VOCs are present in various excreted biological materials (urine, blood, faeces an breath) and their analysis offers a possibility for cancer screening. Some of these VOCs are reversed in the venous blood stream and reach the lung alveoli where some of them are exhaled.

Colorectal cancer (CRC) is one of the commonest tumours and is an important cause of cancer-related mortality. Colonoscopy is the gold standard for the diagnosis of CRC, although its cost prevents its use for mass screening. Furthermore colonoscopy is not well accepted by patients since it is an invasive exam. Screening with fecal immunochemical test (FIT) is associated with a 13-18% CRC-mortality reduction in major randomized studies and is the most widely used non-invasive screening tool, showing fairly good specificity but a high variation in sensitivity (61-91%) and adherence to screening programmes rarely reaches 50-70% of the target population.

Recently the breath analysis has been demonstrated to be a new well accepted and non-invasive tool to detect colorectal cancer.

The purpose of this trial is to compare the reliability of this breath analysis with Immunochemically-based Fecal Occult Blood Test, which is the routinely employed tool for mass screening. A group of subjects adherent to the regional screening program for colorectal cancer prevention, who resulted positive to the FIT, will be enrolled in this study, and will have a breath sampling before undergoing colonoscopy. The predictive ability of the Breath test will be tested in a blind fashion in this selected group of high-risk subjects.

ELIGIBILITY:
Inclusion Criteria:

* Patients with and without positive FIT with a planned colonoscopy
* Patients included in the regional screening program for CRC
* Written informed consent

Exclusion Criteria:

* Pregnancy
* Inflammatory bowel disease
* Bowel prep
* Any psychiatric disease
* Previous (or still present) cancers in other organs

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-05-02 (Actual); Primary Completion 2022-05-02 (Estimated); Study Completion 2022-05-30 (Estimated)

PRIMARY OUTCOMES:
FIT sensitivity | 30 days
  Evaluate the sensitivity of fecal immunochemical test to detect Colorectal cancer patients
Breath analysis sensitivity | 30 days
  Evaluate the sensitivity Breath analysis to detect colorectal cancer patients

CONTACTS AND LOCATIONS:
Overall Officials: Elisabetta Martinelli, MD, Study Chair — Societa Italiana di Chirurgia ColoRettale
Locations (1):
- Dept of Emergency and Organ transplantation, Bari, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Bond A, Greenwood R, Lewis S, Corfe B, Sarkar S, O'Toole P, Rooney P, Burkitt M, Hold G, Probert C. Volatile organic compounds emitted from faeces as a biomarker for colorectal cancer. Aliment Pharmacol Ther. 2019 Apr;49(8):1005-1012. doi: 10.1111/apt.15140. Epub 2019 Mar 3. PMID 30828825
- [Result] Altomare DF, Di Lena M, Porcelli F, Trizio L, Travaglio E, Tutino M, Dragonieri S, Memeo V, de Gennaro G. Exhaled volatile organic compounds identify patients with colorectal cancer. Br J Surg. 2013 Jan;100(1):144-50. doi: 10.1002/bjs.8942. PMID 23212621
- [Result] Stracci F, Zorzi M, Grazzini G. Colorectal cancer screening: tests, strategies, and perspectives. Front Public Health. 2014 Oct 27;2:210. doi: 10.3389/fpubh.2014.00210. eCollection 2014. PMID 25386553
- [Result] Mousavinezhad M, Majdzadeh R, Akbari Sari A, Delavari A, Mohtasham F. The effectiveness of FOBT vs. FIT: A meta-analysis on colorectal cancer screening test. Med J Islam Repub Iran. 2016 May 9;30:366. eCollection 2016. PMID 27493910